CLINICAL TRIAL: NCT02393651
Title: Late LTP-like Plasticity Effects of tDCS in Subacute Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Rick van der Vliet, MSc, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEC-2014-503; NL49887.078.14 (Other: CCMO)
Record Dates: First submitted 2015-03-15; First posted 2015-03-19 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Stroke; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham (Placebo Comparator): Motor training of the affected upper extremity combined with sham tDCS.
  Interventions: Device: tDCS
- tDCS (Experimental): Motor training of the affected upper extremity combined with dual transcranial direct current stimulation (tDCS).
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Late LTP-like plasticity tDCS (2 times per week) for 4 weeks.

SUMMARY:
Rationale: About 80% of stroke patients suffer motor impairments, but current therapies have limited effects on motor recovery. Therefore, investigating new potential therapeutic approaches is crucial. Transcranial Direct Current Stimulation (tDCS) is a form of non-invasive electrical stimulation where a weak current is applied through electrodes over the scalp. This stimulation is known to (1) induce changes in neuronal excitability -which can last up to one day with late LTP-like plasticity protocols in a polarity and site-specific manner, and (2) facilitate motor learning and stroke recovery. So far, several pilot studies have reported beneficial results from tDCS in both subacute and chronic stroke patients, but it's still unclear how tDCS should be repeated over multiple days to optimally enhance recovery and training effects. Using a late LTP-like plasticity protocol could increase effectiveness of standard clinical care rehabilitation sessions and thus enhance the effects of rehabilitation. Therefore, the investigators want to investigate how late LTP-like plasticity tDCS affects rehabilitation in subacute stroke patients. The outcome of this study can provide important guidelines on effective motor therapy during stroke rehabilitation.

Objective: Identify the effect of late LTP-like plasticity on motor rehabilitation during the subacute phase after stroke.

Study design: Double-blinded, randomized between-subjects trials. Study population: Subacute stroke patients. Main study parameters/endpoints: The primary outcome measure is the upper limb motor function during the subacute phase after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subacute stroke (within 1-4 weeks post stroke)
* Acute hemiparesis (Fugl-Meyer Stage < IV) with single thromboembolic non-hemorrhagic infarction documented by a neurologist
* Aged 18-79

Exclusion Criteria:

* Absence of voluntary movement (Fugl-Meyer Stage < III)
* Head injury or the presence of intracranial metal or intracranial lesions
* History of cranial irradiation
* History of epilepsy
* Presence of a pacemaker
* Taking anticonvulsant or neuroleptic medication
* Substance abuse
* Inability to understand instructions

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Upper Extremity Fugl Meyer Assessment | Baseline, 1 week, 2 weeks, 4 weeks and 12 weeks

SECONDARY OUTCOMES:
ARAT | Baseline, 1 week, 2 weeks, 4 weeks and 12 weeks
Hand grip strength | Baseline, 1 week, 2 weeks, 4 weeks and 12 weeks
10-meter walk test | Baseline; 1 week, 2 weeks, 4 weeks and 12 weeks
EuroQol-5D | 12 weeks
Barthel Index | Baseline; 1 week, 2 weeks, 4 weeks and 12 weeks
HADS | Baseline; 4 weeks and 12 weeks
MoCA | Baseline; 4 weeks and 12 weeks
Wong-Baker FACES Pain Rating Scale | Every stimulation session

CONTACTS AND LOCATIONS:
Locations (1):
- Rijndam, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411